CLINICAL TRIAL: NCT02327429
Title: Pilot Test of a Chinese Menu Plan for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Catherine Chan, Professor, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00053775
Record Dates: First submitted 2014-12-18; First posted 2014-12-30 (Estimated); Results first posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A Chinese menu plan for type 2 diabetes (Experimental): All participants will be in the intervention arm for this pilot study
  Interventions: Behavioral: A Chinese menu plan for type 2 diabetes

INTERVENTIONS:
Behavioral: A Chinese menu plan for type 2 diabetes — The intervention is a menu plan, recipes and tips on healthy eating delivered one-on-one between the participant and the facilitator. There will be 4 such one-on-one meetings. The goal is to facilitate behaviour change that results in a healthier diet.

SUMMARY:
In Canada, there is a fast-growing population with diabetes, and the majority of diabetes cases are type 2 diabetes (T2D). Diabetes and its complications, such as cardiovascular diseases, eye disease and foot disease, impair the quality of life and life expectancy.

Chinese are the second largest visible minority in Canada. The diabetes incidence increased much more rapidly in the Canadian population of Chinese origin compared with that of European origin in past decades. Cultural factors are very likely to affect individual behaviour in diabetes treatment. Both international and Canadian diabetes organizations have recognized the importance of taking into account the cultural background and individual preferences in diabetes treatment.

However, there lacks cultural relevant nutritional recommendations or guidelines for Chinese Canadians except some literally translated materials which may not be culturally relevant. In order to fill the gap, the investigators have developed a Chinese menu plan that includes commonly consumed Chinese dishes with nutrients breakdown and cooking tips to provide guidance for patients in their daily meal planning. This menu plan is a cultural translation of the Canadian nutritional guidelines, which is urgently needed among Chinese immigrants with T2D in Edmonton, according to our previous needs assessment.

In this pilot test, the investigators will examine the feasibility and effectiveness of the Chinese menu plan. Twenty Chinese with T2D in Edmonton will be recruited to use the menu plan for 3 consecutive months and relevant indices of T2D will be tested as indicators of effectiveness. Feedback from participants will be obtained through one-on-one interviews and appropriate modifications will be made to the menu plan.

DETAILED DESCRIPTION:
1. Objectives

   The objectives of this study are to assess the feasibility of the Chinese menu plan in Chinese immigrants with type 2 diabetes (T2D), and to assess the effectiveness of the menu plan in terms of nutrient intakes, glycemic control, weight management and other biochemical indices.
2. Background

   2.1 Prevalence of diabetes

   According to Statistics Canada, the diabetes population in 2010 increased by 39.0% compared with that in 2005, while the total population increased by 4.8% in the five years. Diabetes is the sixth leading cause of death in Canada and it brings complications such as cardiovascular, renal, foot and eye diseases, which cause disabilities and reduction in life expectancy. T2D comprises 90% of diabetes population worldwide, and is largely a result of excess body weight and physical inactivity.

   Ethnic Chinese is the second largest visible minority in Canada, and comprises 3.9% and 5.2% of the total population of Canada and of Edmonton, respectively. It has been reported that Chinese Canadians are at high risk of diabetes. This warrants more attention to diabetes management among ethnic Chinese in Canada.

   2.2 Importance of culturally relevant interventions

   Self-care during chronic disease is better facilitated when cultural competence and congruency is incorporated in the management approach. Both international and Canadian guidelines recognize the importance of individualizing treatment based on culture. Chinese Canadians especially the first generations, usually have distinct dietary pattern from the Western diet in terms of food selections and combinations, cooking methods, and the number of dishes per meal, etc. So a general Canadian menu plan is not applicable to ethnic Chinese. Although dietary acculturation happens following immigration, which results in a mixture of traditional and Western diet and cooking techniques in immigrants, traditional diet still takes larger proportion. Diabetes research on Chinese Canadians is scarce and so is Chinese-culture specific nutritional guidelines in Canada. We have developed a culturally relevant menu plan for Chinese Canadians based on the needs assessment and recommendations from Canadian Diabetes Association guidelines and Eating Well with Canada's Food Guide. This pilot study is to test the effectiveness of the menu plan, which can become a practical tool for diabetes self-management in the ethnic Chinese population.
3. Methods and procedures

We will recruit 20 Chinese individuals with T2D in Edmonton to the pilot test. Inclusion criteria are: ≥ 35 years of age; diagnosed with T2D or prediabetes; beginning hemoglobin A1C ≥ 6.0%; treatment with lifestyle, and/or oral hypoglycemic medications or insulin; Chinese origin; able to read and write Chinese or English. Exclusion criteria are: severe gastrointestinal or renal problems that would preclude them eating according to the Nutrition Therapy Guidelines for Diabetes.

3.1 Baseline assessment

Before the 12-week intervention, baseline assessment will be conducted on all participants, including measurement of A1C, height, weight, waist circumference and body composition. Fasting blood samples will be collected for lipid profile measurement. Demographic characteristics, diabetes treatment, self-care activities, physical activity and perceived dietary adherence will be assessed using questionnaires. Participants will three-day food records for dietary intake analysis.

3.2 Adoption

Participants will be asked to follow the menu plan for 12 weeks and keep weekly records of their use of the menu plan. Goal setting will be applied to facilitate adoption. During the first four weeks, the study coordinator will hold one-on-one weekly interviews with each participant to provide feedback and education about the menu plan. Obstacles and strategies will be discussed. During the last eight weeks, only one interview per month will be scheduled to address any problems that participants may have and to help monitor their goal achievement. Participants will be asked to complete another 3-day food record during the last week of the test.

3.3 Final assessment

After study completion, A1C, weight, waist circumference and body composition will be measured within 1 week. A fasting blood sample will be collected to measure lipid profile. Some of the baseline questionnaires including diabetes treatment and perceived dietary adherence will be repeated, and an exit survey will be completed. The final three-day food records will be collected from participants. Focus groups will be conducted to gather information on participants' experiences and perceived benefits of, and barriers and facilitators to following the menu plan. Feedback will be collected as one of the references for possible modification of the menu plan.

3.4 Follow-up

Email or telephone follow-up will be conducted 2 months after study completion to document whether participants continue to use the menu plan. This will be one of the indicators for the long-term feasibility of the menu plan.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 35 years of age;
* diagnosed with T2D or prediabetes;
* baseline hemoglobin A1C ≥ 6.0%;
* treatment with lifestyle, and/or oral hypoglycemic medications or insulin;
* Chinese origin;
* able to read and write Chinese or English

Exclusion Criteria:

* severe gastrointestinal or renal problems that would preclude a diet according to the Nutrition Therapy Guidelines for Diabetes

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Started | 19
Completed | 17
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Program completes only
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 17
Age at Immigration [Mean (Standard Deviation); unit: years] | 45 (19)
Years in North America [Mean (Standard Deviation); unit: years] | 21 (19)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 11 (8)
Acculturation score [Mean (Standard Deviation); unit: units on a scale] — Suinn-Lew Asian Self Identity Acculturation Scale minimum = 1, maximum = 5; lower score indicates lower acculturation
  units on a scale | 1.9 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Energy Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
kcal | -299 (603)

2. Primary Outcome: Change in Carbohydrate Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total energy
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
percentage of total energy | 0.4 (10.3)

3. Primary Outcome: Change in Protein Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total energy
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
percentage of total energy | 1.7 (5.3)

4. Primary Outcome: Change in Total Fat Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total energy
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
percentage of total energy | 0.6 (6.8)

5. Primary Outcome: Change in Saturated Fat Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total energy
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
percentage of total energy | 0.1 (1.9)

6. Primary Outcome: Change in Dietary Fibre Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
grams | 0.8 (13.9)

7. Primary Outcome: Change in Added Sucrose Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of total energy
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
percentage of total energy | 0.2 (1.0)

8. Primary Outcome: Change in Sodium Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
milligrams | -275 (981)

9. Primary Outcome: Change in Calcium Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
milligrams | 124 (341)

10. Primary Outcome: Change in Cholesterol Intake (3-day Food Record)
Description: Intake assessed pre-post intervention using a 3-day food record from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
milligrams | 11 (130)

11. Secondary Outcome: Change in Hemoglobin A1c (A1c)
Description: Hemoglobin A1c measured in capillary blood pre-post intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of A1c in blood
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
% of A1c in blood | -0.13 (0.49)

12. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Body mass index calculated from weight measured pre-post and height measured pre-intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
kg/m2 | -0.4 (0.8)

13. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference measured pre-post intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
cm | -2.0 (2.5)

14. Secondary Outcome: Change in Fasting Triglyceride
Description: Fasting triglyceride measured pre-post intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
mg/dL | -1.2 (88.8)

15. Secondary Outcome: Change in Fasting Total Cholesterol
Description: Fasting total cholesterol measured pre-post intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
mg/dL | -21.4 (28.2)

16. Secondary Outcome: Change in Fasting Low-density Lipoprotein Cholesterol
Description: Low-density lipoprotein cholesterol measured pre-post intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
mg/dL | -18.4 (24.6)

17. Secondary Outcome: Change in Fasting High-density Lipoprotein Cholesterol
Description: Fasting high-density lipoprotein cholesterol measured pre-post intervention from baseline to 3 months
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Number analyzed (Participants) | 17
mg/dL | -2.8 (20.5)

ADVERSE EVENTS:
Time Frame: Total Number of Participants at Risk (e.g., serious and/or other [non-serious] adverse events) were not collected/assessed
Description: Total Number of Participants at Risk (e.g., serious and/or other [non-serious] adverse events) were not collected/assessed. This trial involved working with participants to modify their diets based on nutrition education and a menu plan. Participants were not asked to eat any specific foods, they could modify their diets based on their own preferences; therefore we did not collect information on adverse events since none were anticipated.
Arm/Group | A Chinese Menu Plan for Type 2 Diabetes
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No